## **Document 2: Informed Consent Form**

• **Document Date**: August 1, 2025

o Month: August

o **Day**: 1

**Year**: 2025

• **Document Type**: Informed Consent Form

## • Description:

The Informed Consent Form (ICF) was provided to caregivers of chemotherapy patients participating in the study at Van University Hospital, Turkey. The ICF outlines:

- Study Purpose: To evaluate the impact of a structured educational intervention on caregivers' family health, nutrition, and psychological well-being.
- Procedures: Participation involves completing questionnaires at three time points and, for the intervention group, attending 30–45-minute education sessions.
- o **Risks and Benefits**: Minimal risks (e.g., time commitment); potential benefits include improved health knowledge and well-being.
- Voluntary Participation: Participants can withdraw at any time without consequences.